CLINICAL TRIAL: NCT04986917
Title: Laparoscopic Ventral Hernia Repair with Routine Defect Closure Using Su2ura® Approximation Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anchora Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANC-002
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Ventral Hernia
Keywords: hernia; primary; ventral; laparoscopy; umbilical
MeSH Terms: conditions — Hernia, Ventral; Hernia | interventions — Physical Examination; Vital Signs; Hematologic Tests

STUDY DESIGN:
Intervention Model Description: A total of 60 patients will be recruited to the study. Patients with a primary umbilical hernia under 2 cm will be recruited to the study and the hernia will be repaired with or without mesh according to the PI's decision.
  Eligible patients with a primary or secondary ventral hernia, desiring an elective surgical repair, who amply the inclusion/Exclusion criteria will be offered to participate in the study.
  Study includes 5 visits: Screening, Baseline/Surgery, and 14 days, 3 months, 12months Follow-Ups post-surgery. The actual point of enrollment for each subject is considered the day of surgery. Total study duration is up to 12months post-surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Su2ura® approximation device - study device group (Experimental): Patients with a primary umbilical hernia will be recruited to the study and the hernia will be repaired using the Su2ura® approximation device
  Interventions: Device: Hernia repair surgery using the Su2ura® approximation device; Diagnostic Test: Physical Examination; Diagnostic Test: Vital Signs; Diagnostic Test: Blood Tests; Diagnostic Test: Urine Pregnancy Test; Diagnostic Test: Abdominal Ultrasound imaging; Other: EuraHS-QoL; Other: Visual Analouge Scale (VAS); Diagnostic Test: Clinical evaluation for hernia recurrence and clinical bulging

INTERVENTIONS:
Device: Hernia repair surgery using the Su2ura® approximation device — . The hernia defect will be measured and the Su2ura® approximation device will then be used to close the defect, placing stainless steel implantable anchors threaded on a Polyethylene braided surgical suture.
  Other Names: study device intervention
Diagnostic Test: Physical Examination — All subjects will undergo a standard physical examination by an authorized physician. The physician's evaluation will include diagnosis and documentation of any significant clinical abnormalities or diseases.
Diagnostic Test: Vital Signs — Vital signs include blood pressure, pulse, temperature, body weight and height, body mass index (BMI).
Diagnostic Test: Blood Tests — All subjects will undergo Hematology and Biochemistry blood tests. Blood Hematology test will include a complete CBC. Blood Biochemistry test will include the following measures: Sodium (Na), Potassium (K), Chloride (Cl), Creatinine, Glucose, Urea, Albumin, Calcium total, Alkaline Phosphatase (ALP), ALT, AST, Total Bilirubin, Direct Bilirubin, LDH, Total Protein, Uric Acid, CRP, and Lipid Profile (including Total Cholesterol, HDL, LDL, Triglycerides).
  5 ml of blood (equals to 1 spoon) will be taken for each test.
Diagnostic Test: Urine Pregnancy Test — Urine pregnancy test will be performed during the screening visit (for WOCBP).
Diagnostic Test: Abdominal Ultrasound imaging — All subjects will undergo an abdominal ultrasound (US) imaging at 12 Months visit. The US will be performed to verify an absence of hernia recurrence.
Other: EuraHS-QoL — patients will be asked to fill a questionnaire assessing patient-reported satisfaction and function. questionnaire score range: 0-180; higher score indicates higher pain and discomfort
  Other Names: (hernia-specific European Hernia Society Quality of Life Questionnaire)
Other: Visual Analouge Scale (VAS) — A validated, subjective measure measuring acute and chronic pain. questionnaire score range: 0-10; higher score indicates higher pain level.
Diagnostic Test: Clinical evaluation for hernia recurrence and clinical bulging — The procedure includes:
  1. Clinical examination to determine the presence of hernia recurrence and clinical bulging, in an inconclusive physical exam a radiological imaging will be performed such as US or CT.
  2. SAE's and SADE's evaluation of the seroma.
  3. Taking a photograph of the surgery area without disclosing the subject's identity.

SUMMARY:
Study includes 5 visits: Screening, Baseline/Surgery, and 14 days, 3 months, 12months Follow-Ups post-surgery. The actual point of enrollment for each subject is considered the day of surgery. Total study duration is up to 12 months post-surgery.

Surgery will be performed under general anesthesia. Standard antibiotic prophylaxis will be administered 30 min prior to skin incision. A surgical assistant will be selected by the PI from the surgical staff of the department.

The procedure will involve placement of laparoscopic ports, reduction of the hernia sac, closure of the defect with the Su2ura® approximation device and fixation of mesh with tacks over the closed defect in an IPOM fashion.

Based on surgeon consideration, primary umbilical hernia defects under 2 cm will be repaired with or without mesh.

Study follow-up visits will take place 14 days, 3 months and 12 months post-surgery.

DETAILED DESCRIPTION:
This study will be performed in accordance with the design and specific provisions of this protocol, in accordance with the ethical principles that have their origin in the Declaration of Helsinki, that are consistent with Good Clinical Practice (GCP), Title 21 of the Code of Federal Regulations (21 CFR), part 812 (Investigational Device Exemptions), and the applicable regulatory requirements.

The study is a prospective, multi-center, open study, to evaluate the efficacy and safety of the Su2ura® approximation device.

An abdominal hernia emerges through a preformed or acquired defect of the abdominal wall. The defect may be congenital (primary), acquired as a result of wear and tear (primary), or result from surgery or trauma, where failure of the abdominal wall to heal produces an incisional (non-primary) hernia. Examples of abdominal hernia include epigastric, umbilical and inguinal hernia. Patients may be asymptomatic or complain of a lump or pain. These patients are offered elective surgery. Patients may also present with complications necessitating emergency repair with or without additional resection of compromised viscera.

Ventral hernias are very common and do present a challenge because of the risk of recurrence. Besides the surgeon, these hernias are ideally managed by a dietitian, nurse, and a physical therapist. Patient education has been a very popular topic in literature and hospital settings. Giving patients literature and discussing outcomes with instructions on multiple aspects throughout their encounters has shown to be very effective.

The Su2ura Approximation Device is designed to deploy anchors threaded with stiches to facilitate tissue approximation by eliminating the need for the passing of a needle from one side of the tissue to the other as performed in traditional suturing. Utilizing the anchor feature allows a single action placement of a suture.

The principal investigator from each medical center participated in an appropriate training program. This training included the surgery procedure in an animal. The Principal investigators will train the sub investigators in this procedure. The sponsor will also provide training on the laparoscopic simulator to the principal investigators.

A total of 60 patients will be recruited to the study. Patients with a primary umbilical hernia under 2 cm will be recruited to the study and the hernia will be repaired with or without mesh according to the PI's decision.

Eligible patients with a primary or secondary ventral hernia, desiring an elective surgical repair, who amply the inclusion/Exclusion criteria will be offered to participate in the study.

Study includes 5 visits: Screening, Baseline/Surgery, and 14 days, 3 months, 12months Follow-Ups post-surgery. The actual point of enrollment for each subject is considered the day of surgery. Total study duration is up to 12months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patient desires an elective surgical repair.
3. Patient is able to provide an informed consent.
4. Diagnosis of a primary or secondary ventral hernia, with a fascial defect of width no more than 5 cm width in size on clinical examination or imaging scan.
5. Body mass index (BMI) of 20-40 kg/m2.
6. Candidate for laparoscopic repair based on the operating surgeon's assessment.

Exclusion Criteria:

Exclusion criteria 1. Diagnosis of concomitant abdominal wall defect(s) contiguous with ventral hernia.

2. Patient in need of concomitant non-hernia repair surgical procedure(s). 3. Patient in need of emergent ventral hernia repair for complications such as incarceration, intestinal obstruction or strangulation.

4. The patient desires hernia repair using a technique other than that consistent with the study.

5. Patient has loss of domain as assessed on physical examination or CT scan. 6. Patient has a history of an abdominal aortic aneurysm repair. 7. Patient has a severe co-morbid condition likely to limit survival to less than 2 years.

8. Patient was treated with chemotherapy in the past 6 months. 9. Patient was treated with steroids in the past 6 months. 10. Patient with known collagen disorder. 11. Clean contaminated/contaminated or dirty surgical field. 12. Patient is pregnant or intends to become pregnant during the study period. 13. Patient has ascites on physical examination or CT scan. 14. Patient has liver failure. 15. Patient undergoing dialysis treatment. 16. Patient has a wound-healing disorder. 17. Patient has an untreated coagulation disorder or is on anti-coagulant therapy not managed peri-operatively with the advice or supervision of a hematologist.

18. Patient with autoimmune disorder requiring more than 10 mg of corticosteroid daily.

19. Patient who is immunocompromised (including a diagnosis of HIV/AIDS, organ transplant, or receiving chemo- or radiation therapy.

20. Patient in need of concomitant surgical procedures other than indicated in the protocol as acceptable.

21. Non-compliance with the study protocol. 22. Patient requests to exit the study. 23. Prior radiotherapy. 24. Active malignancy for at least 2 years. 25. Patients has Diastasis recti more than 4cm×4cm size

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Adverse events assesments | up to 30 days
  Overall rate of Serious Adverse Events and serious adverse device effects (SADE) related to study product up to hospital discharge and up to the 30th post-operative day.

SECONDARY OUTCOMES:
Hernia recurrence rate | up to 12 months
  Hernia recurrence rate (Investigator confirmed hernia recurrence on physical examination or imaging).
Patient satisfaction | up to 14 days
  2. Patient satisfaction and function as assessed by the European Hernia Society Quality of life questionnaire (EuraHS-QoL). score range : 0-180 pts; higher score means high pain and discomfort levels.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Hillel Yaffe Medical Center, Hadera, Central District
  - Barzilai Medical Center, Ashkelon, Southern District

IPD SHARING:
Plan to Share IPD: No